CLINICAL TRIAL: NCT05297032
Title: Evaluation of a Computational Model That Predicts the Effects of Quercetin on Metabolic Health Using Biological Age and Other Lipid-related Blood Metrics
Brief Title: Effects of Quercetin on Metabolic Health
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Labs ordering channel is no longer available. Indena (collaborator) opted not to increase funding for an alternative, terminated study.
Sponsor: Thorne HealthTech, Inc (Industry)
Collaborators: Indena S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TRIn-QP01
Record Dates: First submitted 2021-12-09; First posted 2022-03-25 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Quercetin; Lipid Metabolism; Aging
Keywords: Quercetin; Quercetin Phytosome; Quercefit; Sophora japonica; Lipids; LDL; HDL; LDL Particles; Triglycerides; Cholesterol; Metabolic Age; Biological Age; Metabolic Health; Metabolism; Blood Test
MeSH Terms: interventions — Quercetin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Quercetin Phytosome (Experimental): All participants will receive Quercetin Phytosome
  Interventions: Dietary Supplement: Quercetin Phytosome

INTERVENTIONS:
Dietary Supplement: Quercetin Phytosome — All participants will ingest 1 capsule of Quercetin Phytosome (250 mg) three times daily with meals for 90 days.
  Other Names: Quercetin; Quercefit; Sophora japonica extract (flower)

SUMMARY:
Quercetin is a natural flavonoid compound widely found in vegetables, fruits, and nuts. It has a long history of use as a dietary supplement. This study aims to assess results from a computational model suggesting that quercetin may offer novel benefits to metabolic health. Participants will take quercetin (as Quercetin Phytosome, a proprietary formulation with enhanced absorption properties) for 90 days while keeping lifestyle habits consistent throughout to estimate net effects of quercetin as much as possible. Blood samples will be collected at the beginning and end of the study to assess the effects of quercetin supplementation on metabolic health metrics such as LDL cholesterol, blood sugar, liver, kidney and immune function and calculated metabolic age. In addition, questionnaires will be completed to ensure compliance with study requirements and assess potential quercetin benefits in the participants' quality of life. This work will provide a proof-of-concept from a computational model of nutraceutical compounds and proposes a new application of quercetin in support of healthy human metabolism.

DETAILED DESCRIPTION:
Following intake and enrollment steps, including providing consent, and approximately one week before other study activities begin, participants will submit an online questionnaire to collect baseline data about lifestyle factors such as diet, exercise, sleep, stress, and general quality of life. During this period they will also receive the study supplement and schedule their first blood draw at a local-to-them Quest Diagnostics facility. Participants will begin taking the study supplement on the day after their first blood draw. Study dosing consists of one capsule of Quercetin Phytosome (Thorne Research, Inc.; 250 mg) taken three times per day with meals for 90 days. Approximately one week after beginning to take study doses, and bi-weekly thereafter, participants will complete an online questionnaire to monitor lifestyle and quality of life factors. The final questionnaire will be completed on the day of or the day after the last study dose is taken. The day after the last study dose, participants will complete a second blood draw at Quest Diagnostics.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-70 years
* Self-report that, within the past 6 months, a medical professional has informed them of, or a blood test result has shown high-healthy Low Density Lipoprotein (LDL) levels (preferred range, if known: 130-159 mg/dL)

AND 2 or more of the following 4 (values are preferred, if known):

* Low-healthy fasting High Density Lipoprotein (HDL < 50 mg/dL)
* High-healthy fasting Triglycerides (TG 150-199 mg/dL)
* High-healthy fasting Blood Sugar (Glucose 100-126 mg/dL)
* Waist Circumference > 40 in for men or > 35 in for women (this may be self-measured)

Also

* Willing and able to travel to a Quest location for both blood draws
* Willing and able to fast (except water) for 12 hours prior to each blood draw
* Willing and able to comply with the study schedule (+/- 2 days)
* Willing and able to complete online questionnaires
* Willing and able to check email for study-related messages regularly (daily) and to use email as the primary means of communication for non-emergency study-related contact with the study team
* Informed consent to participate in the study discussed and signed
* Willing and able to avoid making changes to diet, sleep, stress, exercise, and other lifestyle factors that may influence the study metrics
* Willing and able to avoid use of the following supplements during the study:

  * Quercetin, Berberine, Red Yeast Rice, Fish Oil, Bergamot Juice Extract, Pantethine, Vitamin D3 dosing over 5,000IU daily, Pterostilbene, Aged Garlic, Phytosterols, Niacin (crystalline/acid, not niacinamide), Meriva/curcumin/turmeric

Exclusion Criteria:

* Individuals who live in NY, NJ, RI, SD, ND, HI, or MD (due to lack of availability of WellnessFX or Quest services)
* Individuals who are currently taking any lipid-lowering medications (including statins) or have taken them within the past 6 months.
* Individuals who are currently taking or have taken any lipid-lowering supplements (including quercetin) consistently in the past 4 weeks. Excluded supplements are products that contain:

  o Berberine, Red Yeast Rice, Fish Oil, Bergamot Juice Extract, Pantethine, Vitamin D3 dosing over 5,000IU daily, Pterostilbene, Aged Garlic, Phytosterols, Niacin (crystalline/acid, not niacinamide), Meriva/curcumin/turmeric
* Diagnosed with metabolic syndrome
* Being treated for hypertension
* Known allergy or sensitivity to any components of the trial's nutritional supplement
* Myocardial infarction, coronary artery bypass grafting, percutaneous transluminal coronary angioplasty, or stent within five years
* Known clinical coronary heart disease symptoms
* Known clinical angina
* History of cerebrovascular accident
* Creatinine > 2.5 mg/dL
* Chronic liver disease with AST, ALT, or alkaline phosphatase over 1.5 times normal
* Known cancer within two years
* Clinical congestive heart failure (systolic or diastolic CHF)
* Type 1 or type 2 diabetes mellitus
* Habitual drinking (cutoff at PI discretion using the following guidelines: 8 or more drinks a week) or being a current smoker/vaping
* Pregnant or nursing
* Women of child-bearing age not using an approved contraceptive
* Planned major surgery during the study (1 week before first blood draw and during the 90-day supplementation)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-09-02 (Actual)

PRIMARY OUTCOMES:
Change in Biological Age score from before (day 0) to after (day 90) supplementation | 90 days
  Quantitative changes before and after intervention in calculated metrics of biological age.
  These metrics are calculated by applying the Klemera-Doubal algorithm to a proprietary set of clinical measures. (Scale for each metric: 0-120) (ref: https://academic.oup.com/biomedgerontology/article/74/Supplement_1/S52/5625183?login=true)
Change in Apolipoprotein B from before (day 0) to after (day 90) supplementation | 90 days
  Quantitative changes before and after intervention in Apolipoprotein B test (Quest Diagnostics 91726) (Scale: mg/dL)
Change in Lipoprotein Fractions from before (day 0) to after (day 90) supplementation | 90 days
  Quantitative changes before and after intervention in Lipoprotein Fractionation, Ion Mobility test (Quest Diagnostics 91604) (Scale: particle number)
Quality of Life scale changes from before (day 0) to after (day 90) supplementation | 90 days
  Quantitative changes in The Quality of Life Scale (Scale: 1-100 as determined by ref: http://www.jstor.org/stable/4034400)

SECONDARY OUTCOMES:
Lifestyle changes from before (day 0) to after (day 90) supplementation | 90 days
  Quantitative changes among any time points in metrics of lifestyle measured by questionnaire.
  Questionnaire metrics and scales:
  Stress: 1-10 (little or none:1, extreme:10) Exercise: 1-10 (little or none:1, extreme:10) Diet: 1-10 (very unhealthy:1, very healthy:10) Sleep: 1-10 (very poor:1, excellent:10)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Phipps, ND, PhD, Principal Investigator — Thorne HealthTech, Inc; Loukia Lili, PhD, Principal Investigator — Thorne HealthTech, Inc
Locations (1):
- This is a remote study - participants will find a commercial lab location near them., Summerville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided